CLINICAL TRIAL: NCT07171879
Title: Partial Extraction Therapy for Facial Contour Preservation, "Old is Gold or Time for Change?" A Randomized Clinical Trial
Brief Title: Pontic Shield and Mineralized Plasmatic Matrix for Ridge Preservation
Acronym: PONTIC-MPM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Soaad Tolba Mohammed Tolba Badawi (Other)
Responsible Party: Sponsor-Investigator, Soaad Tolba Mohammed Tolba Badawi, Lecturer of Oral and Maxillofacial Surgery, Faculty of Dentistry, Mansoura University, Mansoura University
Organization: Mansoura University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R.25.09.22
Record Dates: First submitted 2025-09-06; First posted 2025-09-15 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Alveolar Ridge Preservation
Keywords: Partial extraction therapy; Pontic shield; Mineralized plasmatic matrix (MPM); Socket preservation; Wound healing index
MeSH Terms: interventions — 1-methyl-1-piperidinomethane sulfonate

STUDY DESIGN:
Intervention Model Description: Participants were randomized to one of four groups: extraction alone, extraction with MPM, pontic shield alone, or pontic shield with MPM.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Extraction Only (Active Comparator): Patients receive total tooth extraction in the esthetic maxillary zone without any adjunctive grafting.
  Interventions: Procedure: Tooth Extraction only
- Extraction + MPM (Active Comparator): Patients receive total tooth extraction in the esthetic maxillary zone, followed by grafting with MPM.
  Interventions: Procedure: Extraction + MPM
- Pontic Shield Only (Active Comparator): Patients undergo the pontic shield technique, in which a portion of the buccal root is preserved to maintain ridge contour, without grafting.
  Interventions: Procedure: Pontic Shield Only
- Pontic Shield + MPM (Active Comparator): Patients undergo the pontic shield technique combined with MPM grafting for ridge preservation.
  Interventions: Procedure: Pontic Shield + MPM

INTERVENTIONS:
Procedure: Tooth Extraction only — Conventional atraumatic extraction of the non-restorable maxillary tooth in the esthetic zone without socket preservation procedures.
  Arms: Extraction Only
Procedure: Extraction + MPM — Tooth extraction followed by socket grafting using MPM, prepared from autologous blood combined with xenograft bone particles.
  Arms: Extraction + MPM
Procedure: Pontic Shield Only — Partial extraction therapy using the pontic shield technique, in which the buccal root fragment is preserved to maintain ridge contour, without additional grafting.
  Arms: Pontic Shield Only
Procedure: Pontic Shield + MPM — Pontic shield technique combined with grafting using mineralized plasmatic matrix (MPM) for enhanced ridge preservation and healing.
  Arms: Pontic Shield + MPM

SUMMARY:
This study is testing new methods to preserve the jawbone and gum tissue after removing a damaged front tooth. Normally, when a tooth is taken out, the bone and gums in that area shrink, which can make future dental treatment more difficult and affect appearance. A technique called Partial Extraction Therapy (Pontic Shield Technique) keeps part of the tooth root in place to help maintain the natural shape of the bone and gums. Another method, called Mineralized Plasmatic Matrix (MPM), uses a patient's own blood mixed with bone particles to support healing.

In this randomized clinical trial, 56 patients were assigned to one of four groups:

Group I: Tooth extraction only Group II: Tooth extraction with MPM grafting Group III: Pontic shield technique alone Group IV: Pontic shield technique with MPM grafting The main outcome measured was the amount of bone width preserved, using 3D X-rays (CBCT). Other outcomes included bone height and soft-tissue healing over 4 months.

This research will help determine whether the pontic shield technique, with or without MPM, provides better preservation of bone and gum tissue compared to tooth extraction alone.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years).
* Classified as ASA I (healthy) according to the American Society of Anesthesiologists Physical Status Classification.
* Presence of Type 1 extraction sockets (intact buccal bone and soft tissues).
* Adequate oral hygiene.
* Sufficient inter-arch space for prosthetic rehabilitation.
* Willingness to comply with study protocol and follow-up schedule.

Exclusion Criteria:

* Systemic conditions affecting bone metabolism or wound healing (e.g., uncontrolled diabetes, osteoporosis, immunosuppression).
* History of head and neck radiotherapy or bisphosphonate therapy.
* Acute infection or suppuration at the extraction site.
* Severe periodontal disease.
* Root caries or tooth mobility.
* Buccal bone plate loss due to vertical/horizontal root fractures or advanced periodontitis.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
Alveolar Ridge Width Change | Baseline (pre- or immediate post-extraction) to 4 months.
  Mean changes in alveolar ridge width measured at standardized reference points on cone-beam computed tomography (CBCT) Unit of Measure: millimeters (mm)

SECONDARY OUTCOMES:
Buccal and Palatal Bone Height Change | Baseline to 4 months.
  Change in buccal and palatal bone heights measured on CBCT from baseline to 4 months.
  Unit of Measure: mm
Soft-Tissue Healing (Wound Healing Index, WHI) | 1 week and 4 months post-extraction.
  Clinical soft-tissue healing evaluated using the WHI. Unit of Measure: score on 5-point scale with higher values indicating more favorable wound healing.

CONTACTS AND LOCATIONS:
Overall Officials: Soaad Tolba Badawy, Lecturer, Oral Surgery, MU, Principal Investigator — Mansoura University
Locations (1):
- Faculty of Dentistry, Mansoura University, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No